CLINICAL TRIAL: NCT05001217
Title: Chinese Herbal Medicine Treatment Based on Subgroup Differentiation as Adjunct Therapy for Parkinson's Disease: a Pilot add-on, Randomised, Controlled, Pragmatic Clinical Trial
Brief Title: Chinese Herbal Medicine Treatment as Adjunct Therapy for Parkinson's Disease
Acronym: HERB-PARK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKBU
Record Dates: First submitted 2021-07-07; First posted 2021-08-11 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
Keywords: Chinese medicine; Pragmatic trial; MDS-UPDRS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese herbal medicine treatment plus conventional medication (Experimental): Participants will receive integrated medicine treatment combining Chinese herbal treatment, given in the form of granules, and conventional medication for 32 weeks. Patients will be differentiated into 4 subgroups based on their Chinese medicine pattern, and receive herbal treatment accordingly. An existing clinical pathway will guide the diagnosis and treatment of the Chinese medicine patterns. The four pattern subgroups are as follows:
  1) the "Phlegm-heat stirring Wind" subgroup; 2) the "Spleen-and Kidney-Yang" subgroup; 3) the "Internal Stirring of Yang and Wind" subgroup; and 4) the "Qi deficiency and stasis of Blood" subgroup
  To resemble actual clinical practice, minor adjustment of herbal treatment will be possible and also adhere to the mentioned clinical guideline. The dosage of each herbal drug will follow the instructions of China Pharmacopeia.
  Interventions: Drug: Conventional medication; Drug: Chinese herbal medicine treatment
- Conventional medication (Active Comparator): Conventional medication for Parkinson's disease include levodopa, dopamine agonist, Monoamine oxidase-B inhibitors, Catechol-O-methyltransferase inhibitors, etc.
  Interventions: Drug: Conventional medication

INTERVENTIONS:
Drug: Conventional medication — Levodopa, dopamine agonist, Monoamine oxidase-B inhibitors, Catechol-O-methyltransferase inhibitors, etc.
Drug: Chinese herbal medicine treatment — 1. Huanglian Wendan Decoction
  2. Jin Gui Shen Qi Pill
  3. Liu Wei Di Huang Pill plus Tian Ma Gou Teng Decoction
  4. Bu Yang Huan Wu Decoction
  Arms: Chinese herbal medicine treatment plus conventional medication

SUMMARY:
Background: Parkinson's disease (PD) is a prevalent and debilitating condition. Conventional medications cannot control all symptoms and may inflict adverse effects. A survey reported that Chinese herbal medicine (CHM) is frequently sought. Existing CHM trials were contradictory and often of poor quality due to a lack of methodological rigor. A national clinical guideline was drafted in China with diagnostic criteria and treatment strategy of Chinese medicine (CM) patterns subgroups of PD. The suggested CHM was found to exhibit a neuroprotective effect in in vitro and in vivo studies. This trial aims to preliminarily assess the effect of CHM prescribed based on pattern differentiation on PD symptoms and patients' quality of life, and evaluate the feasibility of the trial design for a future large-scale trial.

Methods: This trial will be a pilot assessor- and data analyst blind, add-on, randomised, controlled, pragmatic clinical trial. 160 PD patients will be recruited and randomised into treatment or control groups in a 1:1 ratio. The trial will be conducted over 32 weeks. PD patients in the treatment group will be stratified into subgroups based on CM pattern and receive CHM accordingly in addition to conventional medication (ConM). The control group will receive ConM only. The primary outcome will be part II of the Movement Disorder Society Sponsored Revision of Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Secondary outcomes will include part and total scores of MDS-UPDRS, domain and total scores of Non-motor symptom scale (NMSS). Adverse events will be monitored by monthly follow-ups and questionnaires. Mixed models will be used to analyse data by Jamovi and R.

Expected outcomes: The success of our trial will show that the pragmatic design with subgroup differentiation is feasible and can produce reliable results. It will also provide preliminary data of the effect of CHM on improving clinical outcomes and quality of PD patients. Data collected will be used to optimize the study design of the future large-scale clinical study.

Ethical clearance: Ethical clearance of this study was given by the Research Ethics Committee of Hong Kong Baptist University (REC/20-21/0206).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with PD according to United Kingdom Parkinson's Disease Society Brain Bank (UKPDBB) diagnostic criteria
2. aged 18 to 80 years old
3. under stable ConM treatment with no alteration of dosage in the past 30 days

Exclusion Criteria:

1. secondary PD or atypical parkinsonian disorder
2. used antidepressants in the previous month
3. with concurrent psychiatric, mood, or other neurological disorders
4. suicidal (with suicidal thoughts in the past year)
5. with concurrent severe disorders, such as cancer and myocardial infarction
6. participation in another Chinese herbal medicine clinical study
7. pregnant or breast-feeding
8. Hoehn and Yahr (H&Y) stage 4 or above
9. liver and renal function derangement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
the Movement Disorder Society Sponsored Revision of Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II | from baseline to week 32
  Assesses the self-reported motor experience of the daily living of Parkinson's patients Scale (Higher the score, the more severe the condition or symptom): 0: Normal, 1: Slight, 2: Mild, 3: Moderate, 4: Severe

SECONDARY OUTCOMES:
Part I, III and IV as well as the total score of MDS-UPDRS | from baseline to week 32
  Comprehensively assesses motor, non motor, and motor complications of Parkinson's patients Scale (Higher the score, the more severe the condition or symptom): Scale: 0: Normal, 1: Slight, 2: Mild, 3: Moderate, 4: Severe
Non-motor symptom scale | from baseline to week 32
  Assesses in details the severity of non motor symptoms of Parkinson's Scale (Higher the score, the more severe the condition or symptom): Severity: 0 = None, 1= Mild (symptoms present but causes little distress or disturbance to patient), 2 = Moderate (some distress or disturbance to patient), 3 = Severe (major source of distress or disturbance to patient); Frequency: 1 = Rarely (<1/wk), 2 = Often (1/wk), 3 = Frequent (several times per week), 4 = Very Frequent (daily or all the time)

CONTACTS AND LOCATIONS:
Overall Officials: Min C Li, PhD, Principal Investigator — School of Chinese medicine, Hong Kong Baptist University
Locations (2):
- Hong Kong (2):
  - Department of Medicine, Queen Elizabeth Hospital, Hong Kong
  - Hong Kong Parkinson's Disease Association, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication, including demographics and characteristics, outcome assessment data, etc
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from baseline to week 32

REFERENCES:
- [Derived] Yuen SCS, Chua KK, Zhong LLD, Chan KW, Chan CKH, Chan KL, Lin Z, Mok V, Lau AY, Li M. Chinese herbal medicine treatment based on subgroup differentiation as adjunct therapy for Parkinson's disease: study protocol of a pilot add-on, randomised, controlled, pragmatic clinical trial. Chin Med. 2022 Jan 24;17(1):16. doi: 10.1186/s13020-022-00572-0. PMID 35073963